CLINICAL TRIAL: NCT06852976
Title: A Phase 2a Proof of Concept Open-Label, Randomized, Controlled Study to Evaluate the Safety and Efficacy of MDI-1228-mesylate Gel Compared With Standard of Care Alone in Patients With Diabetic Foot Ulcers
Acronym: DFU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhuhai Rui-Inno Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPT-1228-101
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Standard of Care for Diabetic Foot Ulcer
  Interventions: Other: Standard of Care Alone
- Treatment Arm (Experimental): MDI-1228-mesylate Gel plus Standard of Care
  Interventions: Drug: 0.75% MDI-1228_mesylate gel plus Standard of Care

INTERVENTIONS:
Drug: 0.75% MDI-1228_mesylate gel plus Standard of Care — Approximately 40 subjects will receive 0.75% MDI-1228_mesylate gel twice daily for 12 weeks.
  Other Names: MDI-1228
  Arms: Treatment Arm
Other: Standard of Care Alone — Approximately 20 subjects will receive the standard of care alone including wound cleaning, debribement and other additional care decided by the healthcare provider.
  Other Names: Standard of Care
  Arms: Control Arm

SUMMARY:
The study will evaluate the treatment effect of MDI-1228-mesylate Gel compared with standard of care alone for the complete healing rate at the end of 12 weeks in participants with diabetic foot ulcers (targeted ulcer). In addition, the proportion of subjects whose target ulcer area is reduced by 50% after 12 weeks of treatment.

DETAILED DESCRIPTION:
The study is targeted to enroll approximately sixty subjects with diabetic foot ulcers. All subjects will be randomized at baseline visits at a 2:1 ratio to either receive the study treatment plus standard of care or standard of care alone.

All subjects who meet inclusion/exclusion criteria will have all ulcers treated; however, only one ulcer, the largest, will be selected as the target ulcer.

Before performing any study procedures, all potential subjects will sign an informed consent form (ICF).

The total study duration is anticipated to be up to 18 weeks, including:

* Up to a 14-day screening period
* Up to 12 weeks study treatment
* Up to 4 weeks of follow-up
* End-of-treatment visit will be performed on the last day of treatment (D84)
* End-of-Study visit will be performed at the follow-up visit (D112)

Wound photography should be dedicated to one study site personnel to control variance.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate and comply with all trial requirements and able to provide signed and dated informed consent prior to initiation of any trial procedures;
2. Male or female 18-75 years;
3. Meet diagnostic criteria for a diabetic ulcer with the presence of at least one target ulcer that meets the characteristics:

   * Located on dorsal or plantar surface of foot or below the knee.
   * Wagner grade 2, ulcerated lesion at or below the knee, without systemic infection.
   * The target ulcer should be the largest, and all each individual ulcers size should be less than 25cm2. All ulcers will be treated the same as the target ulcer.
   * Target ulcers persisted for at least 12 weeks prior to enrollment and have been on standard of care for at least 4 weeks prior to enrollment.
   * There is a minimum 3cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot (post-debridement).

Exclusion Criteria:

1. Allergy to the main components or excipients of MDI-1228_mesylate gel, allergy to JAK inhibitors (tofacitib, baricitinib, ruxolitinib), or individuals with allergic constitution.
2. Skin ulcers or chronic wounds caused by electroshock, chemicals, radioactive material etc.
3. The target ulcer has reduced in size by ≥30% in the last 4 weeks under standard treatment.
4. Those with cancerous ulcers or connective tissue diseases including lupus erythematosus, rheumatoid arthritis, scleroderma, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Drug related treatment emergent adverse events | 1-12 weeks
  Incidence (severity and causality) of any drug related local and systemic treatment emergent adverse events （TEAE） for 12 weeks during the study treatment.
Complete Healing and Time to closure for targeted diabetic foot ulcer | 1-12 weeks
  The proportion of subjects with complete healing of the target ulcer area after 12 weeks of treatment

SECONDARY OUTCOMES:
Ulcer area reduced by 50% | 12 weeks
  The proportion of subjects whose ulcer area was reduced by 50% after 12 weeks of treatment. [The ulcer area will be calculated using a photograph of the ulcer area and PI assessment.]

CONTACTS AND LOCATIONS:
Locations (1):
- Site 001, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No